CLINICAL TRIAL: NCT03497429
Title: A Phase 1, Open-label Study of Niraparib as Single Agent in Patients With Advanced Solid Tumors
Brief Title: A Study of Niraparib as Single Agent in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Niraparib-1001; U1111-1209-0340 (Other: WHO); JapicCTI-183911 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumors
Keywords: Drug Therapy
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: Niraparib 200 mg (Experimental): Niraparib 200 milligrams (mg), capsule, once orally on Days 1 - 21 of each 21-day treatment cycle.
  Interventions: Drug: Niraparib
- Cohort 2: Niraparib 300 mg (Experimental): Niraparib 300 mg, capsule, once orally on Days 1 - 21 of each 21-day treatment cycle.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib capsule

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of Niraparib in Japanese participants with advanced solid tumors.

DETAILED DESCRIPTION:
The drug being tested in this study is called Niraparib. Niraparib is being tested to treat Japanese participants with advanced solid tumors. This study will look at the safety, tolerability and pharmacokinetics of Niraparib administered once daily orally.

The study will enroll approximately 12 participants as a maximum. Participants will be assigned to Cohort 1 (21-day treatment cycle). After that, participants will be assigned to Cohort 2 when safety and tolerability of the 200 mg dose will be demonstrated.

This single-center trial will be conducted in Japan. The overall time to participate in this study is approximately 16 months. Participants will make multiple visits to the clinic with final visit approximately 28 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese male or female participants aged 20 years or older on the day of signing informed consent.
2. Participants must have a cytologically- or histologically-confirmed metastatic or locally advanced solid tumor and have failed or progressed after standard therapy, or for which standard therapy does not exist in the opinion of the investigator.
3. Participants must have Performance Status of less than or equal to (<=) 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale.
4. Participants must have adequate organ function as indicated by the following laboratory values:

   1. Hematology

      * Absolute neutrophil count: greater than or equal to (>=) 1500 per microliter (μL)
      * Platelet count: >=100,000/μL
      * Hemoglobin: >=9 gram per deciliter (g/dL)
   2. Kidney

      - Serum creatinine: <=1.5*institutional upper limit of normal (ULN), OR creatinine clearance of >=50 milliliter per minute (mL/min) (as calculated using the Cockcroft Gault equation or measured using 24-hour urine creatinine clearance) for participants with creatinine levels >=1.5*institutional ULN.
   3. Liver

      * Total bilirubin in serum: <=1.5*ULN (except in participants with Gilbert's syndrome). Participants with Gilbert's syndrome may be enrolled if the participant's direct bilirubin is <=1.5*ULN of the direct bilirubin.
      * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): <=2.5*ULN OR <=5*ULN if participants have liver metastases.
   4. Coagulation (does not pertain to participants receiving anticoagulants)

      * Prothrombin time (PT): <=1.2*ULN
      * Activated partial thromboplastin time (aPTT): <=1.2*ULN
5. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice one highly effective method of contraception and one additional effective (barrier) method at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], condoms only, withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

   Male participants, even if surgically sterilized (ie, vasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug. If the female partner of a male participant is of child bearing potential, it should also be advised to use a highly effective method of contraception, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner], condoms only, withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
6. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Participant who have received chemotherapy, radiotherapy, hormonal or biological therapy within 14 days (within 28 days for anticancer monoclonal antibody, within 42 days for nitrosoureas or mitomycin C) prior to Cycle 1 Day 1. If the participant has residual toxicity from prior chemotherapy treatment, such toxicity must be <=Grade 1 (NOTE: participants with Grade 2 alopecia may qualify for this study). If bevacizumab had been used in the past, all bevacizumab-related toxicities must have resolved. Participants with prostate cancer may have been treated with luteinizing hormone-releasing hormone (LH-RH) analogs.
2. Participants who received a known or putative poly (ADP-ribose) polymerase (PARP) inhibitor or other drugs that may inhibit the PARP, either as part of a clinical trial or as standard of care.
3. Participants who initiated bisphosphonate therapy or are adjusting bisphosphonate dose/regimen within 30 days prior to Cycle 1 Day 1. Participants on a stable bisphosphonate regimen are eligible and may continue the treatment.
4. Treatment with any investigational products within 28 days or 5 half-lives (whichever was longer) before Cycle 1 Day 1.
5. Participants who have symptomatic ascites or a symptomatic pleural effusion. A participant who is treated and clinically stable for these conditions is eligible.
6. Participants with a known primary central nervous system (CNS) tumor.
7. Participants with known CNS metastases and/or carcinomatous meningitis are excluded. However, participants with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for 30 days prior to Cycle 1 Day 1 defined as: (1) no evidence of new or enlarging CNS metastases, (2) off steroids, or (3) on a stable dose and administration of steroids.
8. Participants who have a hypersensitivity to the components of the study drugs or their analogs.
9. Participants who are considered to be at high medical risk due to a serious, uncontrolled disease, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days prior to Cycle 1 Day 1) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, uncontrolled hypertension, or any psychiatric disorder that prohibits obtaining informed consent.
10. Participants who have a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the participant's participation throughout the study period, or study participation is not in the best interest of the participant.
11. Known gastrointestinal (GI) disease or GI surgery that could interfere with the GI absorption of study drug, such as difficulty swallowing capsules and total gastrectomy.
12. Participants who have a psychiatric disorder that may interfere with the conduct of the trial.
13. Participant is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the past year) of drug or alcohol abuse.
14. Participants who are pregnant or breast-feeding, or expecting to conceive or be a father of children within the planned duration of the study.

    NOTE: If a breast-feeding woman discontinue breast-feeding, she may be enrolled in the study.
15. Known human immunodeficiency virus positive.
16. Known hepatitis B surface antigen (HBsAg) positive, or known or suspected active hepatitis C virus (HCV) infection.

NOTE: Participants who are positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antibody (HBsAb) can be enrolled but must have an undetectable hepatitis B virus (HBV) viral load. Participants who have positive hepatitis C virus antibody (HCVAb) must have an undetectable HCV viral load.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites.)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 5 April 2018 to 10 February 2020.
Pre-assignment Details: Japanese participants with advanced solid tumors were enrolled in this dose-escalation study to receive niraparib 200 milligram (mg) in Cohort 1 and niraparib 300 mg in Cohort 2.
Groups:
- Cohort 1: Niraparib 200 mg: Niraparib 200 mg, capsule, orally, once daily, in each 21-day treatment cycle until objective disease progression, unacceptable toxicity or until study discontinuation due to any other reasons.
- Cohort 2: Niraparib 300 mg: Niraparib 300 mg, capsule, orally, once daily, in each 21-day treatment cycle until objective disease progression, unacceptable toxicity or until study discontinuation due to any other reasons.
Period: Overall Study
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Started | 3 | 6
Started | 3 | 6
Completed | 0 | 0
Completed | 0 | 0
Not Completed | 3 | 6
Not completed — Progressive disease | 3 | 4
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (13.75) | 61.3 (12.99) | 58.6 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 6 | 9
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.7 (2.08) | 164.0 (7.64) | 164.9 (6.27)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 65.57 (8.976) | 64.23 (6.575) | 64.68 (6.900)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.56 (2.614) | 23.89 (1.887) | 23.78 (1.990)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status assessed participant's performance status on 5 point scale: 0= Fully active, able to carry on all pre-disease performance without restriction; 1= Restricted in physically strenuous activity but ambulatory, able to carry out work of a light or sedentary nature; 2= Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3= limited self-care; 4= Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead. A higher score indicated greater functional impairment.
  Participants
    0 | 2 | 3 | 5
    1 | 1 | 3 | 4
Diagnosis [Count of Participants; unit: Participants]
  Pancreatic Cancer | 1 | 1 | 2
  Other | 2 | 5 | 7
Prior Surgery/Procedure [Count of Participants; unit: Participants]
  Had prior surgery/procedure | 1 | 3 | 4
  Did not have surgery/procedure | 2 | 3 | 5
Prior Radiation Therapy [Count of Participants; unit: Participants]
  Had prior radiation therapy | 3 | 1 | 4
  Did not have prior radiation therapy | 0 | 5 | 5
Breast Cancer Susceptibility Gene 1 (BRCA1) Mutant [Count of Participants; unit: Participants]
  Had BRCA1 mutant | 0 | 0 | 0
  Did not have BRCA1 mutant | 1 | 1 | 2
  Unknown | 2 | 5 | 7
Breast Cancer Susceptibility Gene 2 (BRCA2) Mutant [Count of Participants; unit: Participants]
  Had BRCA2 mutant | 1 | 1 | 2
  Did not have BRCA2 mutant | 0 | 0 | 0
  Unknown | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), v4.03 and defined as any of the following events occurring during Cycle 1 that were considered by investigator to be related with niraparib: Any Grade 5 or 4 hematologic toxicity, except Grade 4 neutropenia less than (<) 7 days; Grade 3 or 4 neutropenia with fever greater than (>) 38.5 degree Celsius and/or infection requiring antibiotic/anti-fungal treatment; Any Grade 3, 4,or 5 non-hematologic toxicity except: Grade 3 nausea, vomiting, diarrhea/dehydration occurring in setting of inadequate compliance with supportive care and lasting <48 hours, Inadequately treated hypersensitivity reactions, Grade 3 acidosis/alkalosis that responded to intervention by improving to less than or equal to (<=) Grade 2 within 48 hours, Isolated asymptomatic Grade 3 amylase elevation, hypercholesterolemia and hypertriglyceridemia; Any TEAE leading to an interruption of niraparib for >14 days.
Time Frame: Baseline up to Day 21 in Cycle 1 (Cycle length=21 days)
Population: The DLT-evaluable set included participants who had received at least 80 percent (%) of planned doses of niraparib in Cycle 1 (for at least 17 days out of 21 days) unless interrupted by study drug-related toxicities and had sufficient follow-up data considered by sponsor and investigator to determine whether DLT occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: From the first dose of the study drug up to 28 days after the last dose of the study drug (up to Cycle 22 Day 49) (Cycle length =21 days)
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
Participants | 3 | 6

3. Primary Outcome: Number of Participants With Grade 3 or Higher TEAEs
Description: TEAEs were graded as per the NCI-CTCAE version 4.03. As per the NCI-CTCAE, Grade 1 (mild, asymptomatic or mild symptoms); Grade 2 (moderate, minimal, local or noninvasive intervention indicated); Grade 3 (severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated); Grade 4 (life-threatening consequences, urgent intervention indicated); Grade 5 (death related to adverse event [AE]).
Time Frame: as for outcome 2
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
Participants | 1 | 6

4. Primary Outcome: Number of Participants With Serious TEAEs
Time Frame: as for outcome 2
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1

5. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to TEAEs
Time Frame: as for outcome 2
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 2

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Niraparib
Time Frame: Cycle 1 Days 1 and 21: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length =21 days)
Population: The pharmacokinetic (PK) analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 442.9 (195.09) | 529.6 (149.22)
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 4
  Cycle 1 Day 21 | 729.2 (387.50) | 1167 (194.94)

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Niraparib
Time Frame: Cycle 1 Days 1 and 21: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length =21 days)
Population: The PK analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
hours
  Cycle 1 Day 1 | 4.000 [1.52 to 4.07] | 4.035 [2.05 to 10.2]
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 4
  Cycle 1 Day 21 | 3.950 [3.83 to 4.03] | 2.890 [2.88 to 6.00]

8. Secondary Outcome: AUC24：Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours for Niraparib
Time Frame: Cycle 1 Days 1 and 21: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length =21 days)
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
Number analyzed (Participants) | 3 | 6
hour*nanogram per milliliter (h*ng/mL)
  Cycle 1 Day 1 | 4931 (2905.0) | 6270 (2631.2)
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 4
  Cycle 1 Day 21 | 13040 (6493.3) | 19540 (3117.2)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were adverse events that started from the first dose of the study drug up to 28 days after the last dose of the study drug (up to Cycle 22 Day 49) (Cycle length =21 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1: Niraparib 200 mg | Cohort 2: Niraparib 300 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Niraparib 200 mg (N=3) | Cohort 2: Niraparib 300 mg (N=6)
Pyelonephritis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Niraparib 200 mg (N=3) | Cohort 2: Niraparib 300 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1
Platelet count decreased (Investigations) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Alanine aminotransferase increased (Investigations) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 3
Blood creatinine increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03497429/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03497429/SAP_001.pdf